CLINICAL TRIAL: NCT01446198
Title: Clinical Evaluation of the APTIMA® HPV Assay Using the PANTHER™ System
Status: Completed | Type: Observational
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: AHPVPS-US11-003
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Human Papilloma Virus Infection
Keywords: HPV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cervical specimens collected in ThinPrep Pap Test vials containing PreservCyt Solution (Hologic, In., Marlborough, MA) with commercially available collection device or cytobrush/spatula combination may be tested with the HPV Assay either pre- or post-Pap processing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AHPV positive and negative subjects

SUMMARY:
The objective is to establish that APTIMA HPV Assay performance on the PANTHER System is comparable to performance on the TIGRIS System.

DETAILED DESCRIPTION:
The APTIMA HPV Assay is an in vitro nucleic acid amplification test for the qualitative detection of E6/E7 viral messenger RNA (mRNA) from 14 high-risk types of human papillomavirus (HPV) in cervical specimens. The high-risk HPV types detected by the assay include: 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68. The APTIMA HPV Assay does not discriminate between the 14 high-risk types. Cervical specimens collected in ThinPrep Pap Test vials containing PreservCyt® Solution with commercially available collection devices (broom-type device or cytobrush/spatula combination) may be tested with the APTIMA HPV Assay either pre- or post-Pap processing. The assay is used with the TIGRIS System and the PANTHER System.

The objective is to establish that APTIMA HPV Assay performance on the PANTHER System is comparable to performance on the TIGRIS System.

ELIGIBILITY:
Inclusion Criteria:

* the sample had an aliquot with a valid positive or negative APTIMA HPV Assay TIGRIS System result (from testing under protocol 2007HPVASCUS30)
* an aliquot is available and suitable for testing, and
* the sample was randomly selected for inclusion.

Exclusion Criteria:

* sample integrity was compromised (eg, stored under unacceptable conditions)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with AHPV Assay positive results and subjects with AHPV negative results
Sampling Method: Non-Probability Sample
Enrollment: 11816 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
HPV Assay result Agreement between TIGRIS and PANTHER Systems | 1 month
  Percent Positive Agreement: The number of samples with a positive HPV Assay result on TIGRIS and PANTHER divided by the number of samples with a positive HPV Assay result on TIGRIS, multiplied by 100
  Percent Negative Agreement: The number of samples with a negative HPV Assay result on TIGRIS and PANTHER divided by the number of samples with a negative HPV Assay result on TIGRIS, multiplied by 100

CONTACTS AND LOCATIONS:
Overall Officials: Tadd S Lazarus, M.D., Study Director — Gen-Probe, Incorporated
Locations (3):
- United States (3):
  - Gen-Probe Incorporated, San Diego, California
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - LabCorp Corporation of America, Burlington, North Carolina